CLINICAL TRIAL: NCT06329960
Title: Efficacy of Ultrasound-guided Dorsal Scapular Nerve Injection Combined With Rhomboideus Muscle Needle Release
Brief Title: Dorsal Scapular Nerve Injection Combined With Muscle Needle Release
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Zhu Jiaan, Chairman, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024PHB019-001(3)
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Dorsal Scapular Nerve Entrapment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Ultrasound-guided dorsal scapular nerve injection combined with needle release of major and minor rhomboideus
  Interventions: Other: Ultrasound-guided injection combined with needle release

INTERVENTIONS:
Other: Ultrasound-guided injection combined with needle release — Ultrasound-guided PIT using D5W HD for dorsal scapular nerve combined with needle release of major and minor rhomboideus

SUMMARY:
Ultrasound-guided perineural injection (PIT) of 5% dextrose (D5W) hydrodissection has been widely used in the treatment of peripheral entrapment neuropathies. However, there are few studies investigating the efficacy of PIT using D5W HD for dorsal scapular nerve (DSN) entrapment. Generally, the DSN entrapment causes the stiffness of the major and minor rhomboideus(2). In clinical practice, the investigators observed that ultrasound-guided PIT using D5W HD combined with needle release of major and minor rhomboideus significantly relieved the pain of scapular region. Therefore, the investigators aimed to evaluate the 6-month efficacy of this procedure for the participants with DSN entrapment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with DSN entrapment confirmed by electrophysiological study;
* age 18-80 years;
* patients who were irresponsive to conservative treatment;
* symptoms persisted for more than 3 months.

Exclusion Criteria:

* pregnancy
* DSN entrapment caused by trauma, surgery or occupying lesions of DSN;
* concurrent presence of rheumatic immune diseases, hypothyroidism, or diabetes mellitus;
* C5/6 lumbar radiculopathy;
* previous history of local injection or surgery for DSN entrapment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
visual analogue scale (VAS) | before treatment, as well as 1, 3, 6 months post treatment
  VAS is the most common tool to evaluate discomfort for patients with peripheral entrapment neuropathies, with scores ranging from 0 (no pain) to 10 (intolerant pain)

CONTACTS AND LOCATIONS:
Overall Officials: Jiaan Zhu, Principal Investigator — Peking University People's Hospital
Locations (1):
- Jiaan Zhu, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lam KHS, Wu YT, Reeves KD, Galluccio F, Allam AE, Peng PWH. Ultrasound-Guided Interventions for Carpal Tunnel Syndrome: A Systematic Review and Meta-Analyses. Diagnostics (Basel). 2023 Mar 16;13(6):1138. doi: 10.3390/diagnostics13061138. PMID 36980446
- [Background] Muir B. Dorsal scapular nerve neuropathy: a narrative review of the literature. J Can Chiropr Assoc. 2017 Aug;61(2):128-144. PMID 28928496